CLINICAL TRIAL: NCT04302792
Title: Oncofood: New Food Solutions for Cancer Patients
Brief Title: New Food Solutions for Cancer Patients
Acronym: Oncofood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: AZTI Spain (Unknown); Maspex Poland (Unknown); Natural Machines Spain (Unknown); University of Warsaw (Other)
Responsible Party: Principal Investigator, Stella Lignou, Lecturer in Sensory and Consumer Science, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Oncofood - 20139
Record Dates: First submitted 2020-02-28; First posted 2020-03-10 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Cancer Patients; Taste Disorders; Food Selection
Keywords: taste & smell alterations; texture-modified foods; taste-optimised foods; cancer patients
MeSH Terms: conditions — Taste Disorders; Food Preferences

STUDY DESIGN:
Intervention Model Description: This is a 3 stage study design. The first stage will be a qualitative part with interviews and focus group sessions. In the second and third stages participants will evaluate food products. The second and third stages of the study will be conducted single blind as it is not feasible to blind the researcher.
Who Masked: Participant
Masking Description: All samples provided to the participant are labelled with 3 digit random codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1: Interviews and focus group sessions (No Intervention): Group A: Cancer patients (requiring or have required texture-modified foods and/or experiencing or have experienced taste&smell alterations in the last 12 months) will be required to attend a one-hour online interview.
  Group B: Relatives of cancer patients (requiring texture-modified foods and/or experiencing taste&smell alterations) will be required to attend a 2-hour online focus group session.
  Group C: Healthcare professionals with a minimum of a year's experience with oncological patients that require texture-modified foods and/or have taste & smell alteration will be required to attend a 2-hour online focus group session.
  A food diary will be given to Group A and B to complete for 7-days prior to their session. Topics to be discussed during the interview and the focus group sessions will include the food requirements of cancer patients, the barriers of the current food products, possible solutions to these requirements if any and their expectations towards new food solutions.
- Stage 2: Texture-modified foods for cancer patients (Experimental): The study will involve conducting a tasting trial over a 2-weeks period where participants will be required to consume a maximum of three 3D printed texture-modified food based on the findings from Stage 1 and evaluate the food product by completing a structured questionnaire. Key questions areas covered by the questionnaire include appetite, sensory characteristics of the product (taste, flavour, mouthfeel/texture and smell), liking and acceptability, purchase intent and best place to buy the products; questions will involve rating scales as well as qualitative comments.
  Interventions: Behavioral: Texture-modified foods for cancer patients (Stage 2)
- Stage 3: Taste-optimised foods for cancer patients (Experimental): The study will involve conducting a home test over a one-month period where participants will be required to consume taste-optimised products based on the findings from Stage 1 and evaluate the food product by completing a structured questionnaire. Key questions areas covered by the questionnaire include appetite, sensory characteristics of the product (taste, flavour, mouthfeel/texture and smell), liking and acceptability, purchase intent and best place to buy the products; questions will involve rating scales as well as qualitative comments.
  Interventions: Behavioral: Taste-optimised foods for cancer patients (Stage 3)

INTERVENTIONS:
Behavioral: Texture-modified foods for cancer patients (Stage 2) — Participants (cancer patients that require texture-modified foods) will be expected to evaluate a maximum of three meals over a 2-weeks period.
  Arms: Stage 2: Texture-modified foods for cancer patients
Behavioral: Taste-optimised foods for cancer patients (Stage 3) — Participants (cancer patients with taste & smell alterations) will be expected to evaluate three foods at home over a period of one month.
  Arms: Stage 3: Taste-optimised foods for cancer patients

SUMMARY:
The ONCOFOOD project aims to design and develop new innovative food solutions for cancer patients, taking into account not only their nutritional requirements but also their sensory changes, promoting eating pleasure and preventing malnutrition. Research involving cancer patients but also their families and health care professionals is a key element of this approach to ensure the success of the developed products for the target group.

DETAILED DESCRIPTION:
The study will be divided into three stages: in Stage 1, individual interviews will be conducted with present and past cancer patients, focus groups with families/care givers of cancer patients and health care professionals (cancer specialist nurses, clinical and medical oncologists, speech and language therapists, dietitians, oncology social workers and counselors). The interviews will help collect data and gain understanding on the needs of cancer patients, barriers to current food proposals and expectations from new solutions. In subsequent stages, semi-quantitative studies will be conducted with cancer patients that require texture-modified foods (Stage 2) and patients with taste & smell alterations (Stage 3). Patients will be required to evaluate texture-modified products (developed using 3D food printing technology) and taste-optimised products (i.e. soups, mousses, fruit and vegetable beverages, dairy desserts and seasonings) developed based on the results obtained from Stage 1 above.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 1

   1. Group A - Patients

      * Adults 18-65 years old.
      * Currently undergoing oncological treatment or have undergone oncological treatment in the last 12 months.
      * Patients that require or have required texture-modified foods and/ or experience or have experienced taste & smell alterations in the last 12 months.
   2. Group B - Relatives and caregivers

      * Over 18 years old.
      * Relative or caregiver of an adult oncological patient (that require texture-modified foods and/ or experience taste & smell alterations).
      * Living/caring for someone that is currently undergoing or have undergone oncological treatment.
      * Participates actively in cooking and buying food for a household of which the person currently undergoing oncological treatment is a member.
   3. Group C - Healthcare professionals

      * Dietitians, speech and language therapists, medical/clinical oncologists, cancer specialist nurses, and oncology social workers and counselors.
      * Minimum of a year's experience with oncological patients that require texture-modified foods and/or having taste & smell alterations.
2. Stage 2

   * Adults 18-65 years old.
   * Currently undergoing oncological treatment or have undergone oncological treatment in the last 12 months and require or have required texture-modified foods in the last 12 months.
   * Individuals without dietary allergies or intolerances to the foods that will be tested in the study.
3. Stage 3

   * Adults 18-65 years old.
   * Currently undergoing oncological treatment or have undergone oncological treatment in the last 12 months and are experiencing or have experienced taste & smell alterations in the last 12 months.
   * Individuals without dietary allergies or intolerances to the foods that will be tested in the study.

Exclusion Criteria:

* Individuals below 18 years old will be excluded from the study.
* Individuals with dietary intolerances or allergies to the foods that will be tested in the study (Stages 2 and 3 only).
* Individuals who do not have the ability or capacity to consent.
* Individuals who are nil by mouth or have nasal gastric tubes of other feeding tubes inserted.
* Individuals who need modified solid and liquid diets due to problems with swallowing (Stage 3 only).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of developed texture-modified food 1 | 1 hour on Stage 2 visit day 1
  Acceptability of texture-modified food 1 using a questionnaire. Participants will be asked to rate their liking of appearance, aroma, taste, texture and overall using a 9-point hedonic scale where 1 is "dislike extremely" and 9 is "like extremely". They will also be asked to indicate their preference in comparison to usual products using a 5-point scale where 1 is "I much preferred this product to my usual products" and 5 is "I much prefer my usual products to this one". They will be asked to indicate whether they would buy this product using a 5-point scale where 1 is "definitely would buy" and 5 is "definitely would not buy".
Acceptability of developed texture-modified food 2 | 1 hour on Stage 2 visit day 2
  Acceptability of texture-modified food 2 using a questionnaire. Participants will be asked to rate their liking of appearance, aroma, taste, texture and overall using a 9-point hedonic scale where 1 is "dislike extremely" and 9 is "like extremely". They will also be asked to indicate their preference in comparison to usual products using a 5-point scale where 1 is "I much preferred this product to my usual products" and 5 is "I much prefer my usual products to this one". They will be asked to indicate whether they would buy this product using a 5-point scale where 1 is "definitely would buy" and 5 is "definitely would not buy".
Acceptability of developed texture-modified food 3 | 1 hour on Stage 2 visit day 3
  Acceptability of texture-modified food 3 using a questionnaire. Participants will be asked to rate their liking of appearance, aroma, taste, texture and overall using a 9-point hedonic scale where 1 is "dislike extremely" and 9 is "like extremely". They will also be asked to indicate their preference in comparison to usual products using a 5-point scale where 1 is "I much preferred this product to my usual products" and 5 is "I much prefer my usual products to this one". They will be asked to indicate whether they would buy this product using a 5-point scale where 1 is "definitely would buy" and 5 is "definitely would not buy".
Acceptability of developed taste-optimised food 1 | 1 hour on Stage 3 visit day 1
  Acceptability of taste-optimised food 1 using a questionnaire. Participants will be asked to rate their liking of appearance, aroma, taste, texture and overall using a 9-point hedonic scale where 1 is "dislike extremely" and 9 is "like extremely". They will also be asked to indicate their preference in comparison to usual products using a 5-point scale where 1 is "I much preferred this product to my usual products" and 5 is "I much prefer my usual products to this one". They will be asked to indicate whether they would buy this product using a 5-point scale where 1 is "definitely would buy" and 5 is "definitely would not buy".
Acceptability of developed taste-optimised food 2 | 1 hour on Stage 3 visit day 2
  Acceptability of taste-optimised food 2 using a questionnaire. Participants will be asked to rate their liking of appearance, aroma, taste, texture and overall using a 9-point hedonic scale where 1 is "dislike extremely" and 9 is "like extremely". They will also be asked to indicate their preference in comparison to usual products using a 5-point scale where 1 is "I much preferred this product to my usual products" and 5 is "I much prefer my usual products to this one". They will be asked to indicate whether they would buy this product using a 5-point scale where 1 is "definitely would buy" and 5 is "definitely would not buy".
Acceptability of developed taste-optimised food 3 | 1 hour on Stage 3 visit day 3
  Acceptability of taste-optimised food 3 using a questionnaire. Participants will be asked to rate their liking of appearance, aroma, taste, texture and overall using a 9-point hedonic scale where 1 is "dislike extremely" and 9 is "like extremely". They will also be asked to indicate their preference in comparison to usual products using a 5-point scale where 1 is "I much preferred this product to my usual products" and 5 is "I much prefer my usual products to this one". They will be asked to indicate whether they would buy this product using a 5-point scale where 1 is "definitely would buy" and 5 is "definitely would not buy".

SECONDARY OUTCOMES:
Food diary | 7 consecutive days
  Record of all that is eaten or drunk and any problems encountered during/after eating from cancer patients and relatives/caregivers of cancer patients.
Interviews | 1 hour session on Stage 1 visit day 1
  Discussion on food related issues faced by cancer patients requiring texture-modified diets / having taste & smell alterations via interviews.
Focus group | 2 hour session on Stage 1 visit day 2
  Discussion on food related issues faced by cancer patients requiring texture-modified diets / having taste & smell alterations with relatives/caregivers of cancer patients via a focus group session.
Focus group | 2 hour session on Stage 1 visit day 3
  Discussion on food related issues faced by cancer patients requiring texture-modified diets / having taste & smell alterations with healthcare professionals of cancer patients via a focus group session.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Lignou, PhD, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Tueros I, Uriarte M. Innovative food products for cancer patients: future directions. J Sci Food Agric. 2018 Mar;98(5):1647-1652. doi: 10.1002/jsfa.8789. Epub 2017 Dec 6. PMID 29168190
- [Background] Wickham RS, Rehwaldt M, Kefer C, Shott S, Abbas K, Glynn-Tucker E, Potter C, Blendowski C. Taste changes experienced by patients receiving chemotherapy. Oncol Nurs Forum. 1999 May;26(4):697-706. PMID 10337648
- [Background] Lovell SJ, Wong HB, Loh KS, Ngo RY, Wilson JA. Impact of dysphagia on quality-of-life in nasopharyngeal carcinoma. Head Neck. 2005 Oct;27(10):864-72. doi: 10.1002/hed.20250. PMID 16114007
- [Background] Amezaga J, Alfaro B, Rios Y, Larraioz A, Ugartemendia G, Urruticoechea A, Tueros I. Assessing taste and smell alterations in cancer patients undergoing chemotherapy according to treatment. Support Care Cancer. 2018 Dec;26(12):4077-4086. doi: 10.1007/s00520-018-4277-z. Epub 2018 May 31. PMID 29855774